CLINICAL TRIAL: NCT03945136
Title: Implementation of Brief Dynamic Interpersonal Therapy at the VA
Acronym: DIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: VA New York Harbor Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cory K. Chen, PhD, Director - Psychotherapy Research and Development Program, VA New York Harbor Healthcare System
Other Study IDs: VANYHH
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Depression; Anxiety
Keywords: veterans; depression; anxiety; psychodynamic; psychotherapy; treatment
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Dynamic Interpersonal Therapy — Dynamic Interpersonal Therapy is a time-limited, manualized, interpersonal and affect-focused psychodynamic treatment that is frequently used to target depression and anxiety.

SUMMARY:
The goal of the proposed project is to collect data from clinician files and the electronic medical record to describe the clinical implementation of Brief Dynamic Interpersonal Therapy (DIT), an individual psychotherapy for depression and anxiety, at the VA through psychology staff and trainees between 2012-present.

DETAILED DESCRIPTION:
The goal of the proposed project is to collect data from clinician files and the electronic medical record to describe the clinical implementation of Brief Dynamic Interpersonal Therapy (DIT), an individual psychotherapy for depression and anxiety, at the VA through psychology staff and trainees between 2012-present. The study will collect data on patient characteristics (e.g. demographics, diagnoses, reasons for referral, etc.), attendance, and treatment outcome of depression, anxiety and psychosocial functioning to evaluate and describe the feasibility of implementing DIT at the VA.

Medical records of veterans who were provided with DIT treatment between 2012-present will be reviewed and data on patient characteristics (which will include demographic information, diagnoses, reasons for referral, etc.), treatment compliance, and treatment outcome as measured by changes in depression, anxiety, and psychosocial functioning during the treatment period and up to the present will be collected. The investigators estimate that approximately 100 Veterans have been offered and/or provided DIT since 2012 by psychology trainees and staff. This study will provide preliminary data on the feasibility of implementing DIT treatment at the VA. The first trial of DIT for MDD in the VHA is currently being conducted by the PI and the information from the retrospective chart review would help to provide additional data as part of a proposal for a larger scale RCT of DIT.

ELIGIBILITY:
Inclusion Criteria:

- receive DIT treatment at VANYHHS between 2012-present

Exclusion Criteria:

- was not referred for, or did not receive at least 1 DIT session at VANYHHS between 2012-present

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans that have received DIT treatment for clinically indicated depression and/or anxiety at VANYHHS (Manhattan) between 2012 to present.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-03-15 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Total score collected at each weekly session of DIT, up to 16 weeks.; Scale: 0-4: Minimal depression; 5-9: Mild depression; 10-14: Moderate Depression; 15-19: Moderately Severe Depression; 20-27: Severe Depression
  The PHQ-9 is used to assess depressive symptom severity in patients.
Generalized Anxiety Disorder Scale - 7 Item (GAD-7) | Total score collected at each weekly session of DIT, up to 16 weeks. Scale: 0-5: Mild Anxiety; 6-10: Moderate Anxiety; 11-15: Severe Anxiety
  The GAD-7 is used to assess anxiety symptom severity in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Cory K Chen, PhD, Principal Investigator — VA New York Harbor Healthcare System
Locations (1):
- VA New York Harbor Healthcare System, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No